CLINICAL TRIAL: NCT03195777
Title: Novel PET/CT and Treatment Strategies to Reduce PTS Following DVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Tawakol, Interim Director, Nuclear Cardiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017P000808
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Deep Venous Thrombosis; Post-thrombotic Syndrome
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: This study is a one-center observational study examining DVT with FDG- PET/CT. 80 individuals with DVT will be imaged with PET/CT and followed for development of PTS
Masking Description: Investigators who are analyzing images will be blinded to all clinical data, including clinical follow-up data to determine PTS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm: Observation after Imaging (Experimental): This is a single-arm study, where subjects will be monitored for development of PTS after baseline non-invasive imaging with FDG PET/CT. The experimental interventIon is the PET/CT imaging.
  Interventions: Device: PET/CT

INTERVENTIONS:
Device: PET/CT — PET/CT imaging will be performed (with fluorodeoxyglucose, [FDG] as a tracer). Thereafter, subjects will be monitored for development of PTS. We will then assess the ability of PET/CT top predict the subsequent development of PTS.

SUMMARY:
The goal of this study is to develop strategies that will improve outcomes for patients with deep vein thrombosis (DVT), using in vivo FDG-PET inflammation imaging to better predict the development of the post-thrombotic syndrome (PTS). New approaches are needed to improve the outcomes of patients with DVT, a disease that affects up to 600,000 patients per year in the US alone. DVT acutely places patients at risk of death from pulmonary embolism and causes 50,000 deaths annually in the US. Moreover, up to 30-50% of patients will develop PTS, an illness characterized by inflammation-driven fibrotic vein wall injury, and persistent thrombus obstruction. PTS occurs despite anticoagulant therapy, and produces chronic disability from leg pain, heaviness, edema, skin pigmentation, and ulcers; some patients may even require amputation. PTS impairs quality of life to the same extent as chronic obstructive pulmonary disease or diabetes. Therefore new diagnostic insights into PTS are urgently needed.

There are several major challenges to improve outcomes in PTS: A) Limited in vivo knowledge regarding inflammation and the development of PTS; B) L Lack of predictive approaches to identify patients at high risk for PTS that will preferentially benefit from novel therapies. Recently, our laboratories have harnessed FDG-PET molecular imaging to illuminate DVT inflammation in vivo, and to provide a new strategy to diagnose recurrent DVT, a vexing clinical problem (Hara et al. Circulation 2014). We now propose to further develop FDG-PET to improve outcomes in DVT and PTS.

The objective of this application is to develop FDG-PET as an inflammation imaging approach to assess DVT inflammation and predict risk of developing PTS in human subjects;

Hypothesis 1A: Inflammatory activity in DVT (quantified acutely, using FDG-PET imaging within 0-7 days after DVT) will predict PTS incidence (primary) and severity (secondary) within a 24 month follow-up period.

Hypothesis 1B: Inflammatory activity in DVTs (quantified sub-acutely, using FDG-PET imaging within 21-28 days after DVT), will predict PTS incidence and severity.

Eighty patients with DVT will be imaged using FDG-PET/CT acutely (0-7 days of DVT diagnosis), and sub-acutely (21-28 days after diagnosis). Subjects will be evaluated repeatedly for up to 2 years to detect clinical evidence of PTS (Villalta score), ultrasound findings for structural venous injury, and soluble biomarkers of systemic inflammation. Subsequently, we will evaluate the relationship between FDG DVT activity and the development of PTS.

DETAILED DESCRIPTION:
This study is a one-center observational study examining DVT with PET/CT. 80 individuals with recent deep venous thrombosis (DVT) will be recruited from MGH. Imaging and clinical evaluation will be performed to look for predictors of a major complication of DVT: the post-thrombotic syndrome (PTS)

There are 5 visits to attend. The imaging visits will last 2-3 hours. The clinical evaluation visits will last 1-2 hours.

1. Screening - This visit will take place after initial DVT (deep venous thrombosis) diagnosis. It will involve clinical assessments and blood labs, to determine subject eligibility. If an ultrasound was not performed at the time of DVT diagnosis, an ultrasound should be performed.
2. Visit 1 (0-7 days after DVT diagnosis) - Imaging Visit 1 - At this visit, patients will receive a positron-emission tomography/ computed tomography (PET/CT) scan, and contrast-enhanced CT of the lower extremity (CTA) and will have blood labs drawn.
3. Visit 2 (21-28 days after DVT diagnosis) - Imaging Visit 2 - At this visit, patients will receive a PET/CT scan and will have blood labs drawn.
4. Visit 3 (6 months after DVT diagnosis) - Clinical Evaluation - At this visit, patients will meet to evaluate symptoms of DVT and PTS. Blood labs will be drawn. An ultrasound will be performed as well.
5. Visit 4 (24 months after DVT diagnosis OR time of PTS diagnosis) - Clinical Evaluation - At this visit, patients will meet to evaluate symptoms of DVT and PTS. Blood labs will be drawn. An ultrasound will be performed as well.

ELIGIBILITY:
Inclusion Criteria:

* Age above 30
* Patient presents with a first symptomatic, proximal DVT (with or without concurrent distal DVT or pulmonary embolism).

Exclusion Criteria:

* Patient has May-Thurner syndrome
* Patient has an expected life span of < 6 months
* Patient can't receive anticoagulation therapy
* Patient received thrombolytic therapy for the initial treatment of acute DVT
* Patient has DVT signs of symptoms that occur more than 1 week prior to presentation, as assessed by clinical history
* Renal dysfunction (Serum creatinine > 1.5 mg/ml or estimated creatinine clearance < 60 ml/min)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-06-08 (Actual)

PRIMARY OUTCOMES:
PTS incidence | 24 month follow-up period
  Incidence of PTS (by Villalta score of ≥5) at any time during 24 months of observation after diagnosis of first proximal DVT

SECONDARY OUTCOMES:
PTS severity | 24 month follow-up period
  Maximal severity of PTS (by Villalta score) during 24 month observation

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hara T, Truelove J, Tawakol A, Wojtkiewicz GR, Hucker WJ, MacNabb MH, Brownell AL, Jokivarsi K, Kessinger CW, Jaff MR, Henke PK, Weissleder R, Jaffer FA. 18F-fluorodeoxyglucose positron emission tomography/computed tomography enables the detection of recurrent same-site deep vein thrombosis by illuminating recently formed, neutrophil-rich thrombus. Circulation. 2014 Sep 23;130(13):1044-52. doi: 10.1161/CIRCULATIONAHA.114.008902. Epub 2014 Jul 28. PMID 25070665